CLINICAL TRIAL: NCT03562975
Title: A Single-center Prospective Measurement of Upper Extremity Function in Multiple Sclerosis Patients With Advanced Disability Treated With Ocrevus™
Brief Title: Upper Extremity Function in Multiple Sclerosis Patients With Advanced Disability Treated With Ocrevus
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCRE-UP
Record Dates: First submitted 2018-05-23; First posted 2018-06-20 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Pathologic Processes; Demyelinating Diseases; Nervous System Diseases; Autoimmune Diseases; Immune System Diseases; Primary Progressive Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Pathologic Processes; Demyelinating Diseases; Nervous System Diseases; Autoimmune Diseases; Immune System Diseases; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab is a humanized anti-CD20 monoclonal antibody. It targets CD20 marker on B lymphocytes and hence is an immunosuppressive drug candidate. Ocrelizumab binds to an epitope that overlaps with the epitope to which rituximab binds
  Other Names: Ocrevus

SUMMARY:
The investigators are measuring the effectiveness of Ocrevus™ in helping patients with hand or arm weakness, especially if posed by a more advanced MS patient than those included in the clinical trials.

DETAILED DESCRIPTION:
Ocrevus™ is the first FDA approved disease-modifying treatment for primary progressive multiple sclerosis (PPMS) as well as relapsing MS. In the clinical trials considered by the FDA (OPERA I/II, ORATORIO), the highest Expanded Disability Status Scale (EDSS) included in the participants was 5.5 (OPERA I/II) and 6.5 (ORATORIO). The EDSS score is heavily weighted on walking ability and is not a useful measurement for UE function. The primary endpoint in the primary progressive MS trial with Ocrevus™ was EDSS and in the relapsing MS studies, EDSS was used as a secondary endpoint. The Multiple Sclerosis Functional Composite (MSFC) score (Z score), a composite of quantitative measure of walking speed, upper limb coordinated movement (9 Hole Peg Test/9HPT) and cognitive function, was obtained as a secondary clinical measure with scores being favorably higher in patients treated with Ocrevus™ (OPERA I/II).The z score, however, is not very useful in delineating which of the three clinical functions was maintained or showed less progression given that three domains are included in the score. Data presented recently from the Oratorio trial analyzed the intention to treat population of PPMS patients and the subgroups of patients with upper extremity functional impairment using the 9HPT; results demonstrated reduction in risk of clinical progression in upper extremity disability in patients treated with Ocrevus compared to placebo. There was improvement in the change from baseline to week 120 in 9HPT time in treated patients. Abnormal baseline 9HPT was defined as >25 seconds and upper extremities were defined as "better hand" and "worse hand", each individually tested, with clinical progression determined at 12 and 24 weeks in 3 sub-categories of progression: lengthened time of 9HPT >15%, >20% and 25%.

In this study, investigators aim to not only replicate the results in the Oratorio trial with upper extremity dysfunction, but also widen the spectrum of patients that may benefit (given an expanded MS population of patients, not exclusive to PPMS and widen the It is anticipated that by using a test that better emulates activities of daily life performed with the upper extremity, such as the TEMPA (Test d'Evaluation de la performance des membres Superieurs e Personnes Agees ) more real life application of the benefits of receiving treatment with Ocrevus will be obtained, and it is anticipated that patients can maintain the function they have or potentially improve function.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent and any authorizations required by local law (e.g., Protected Health Information [PHI])
* Aged 18-70 at the time of informed consent
* Must have a relapsing or progressive form of MS
* Plan to begin Ocrevus™ treatment but have not actually had first treatment yet
* Male subjects and female subjects of child-bearing potential (including female subjects who are not post-menopausal for at least 1 year) must be willing to practice effective contraception (as defined by the investigator) during the study and be willing and able to continue contraception for 6 months after their last dose of study treatment
* EDSS 4.0-8.0
* UE weakness in at least one limb, defined as grade 4/5 in ≥ 2 muscles per limb
* Muscle weakness must be primarily related to MS
* Joint range of motion must be within functional limits
* Patient must be able to perform 9HPT and TEMPA tests with at least one limb

Exclusion Criteria:

* Prior treatment with Ocrevus™ (Cannot already be on Ocrevus prior to joining the study)
* Severe weakness in bilateral upper limbs causing complete loss of function
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity
* Female subjects considering becoming pregnant while in the study
* Female subjects who are currently pregnant or breast-feeding
* Unwillingness or inability to comply with the requirements of the protocol including the presence of any conditional (physical, mental or social) that is likely to affect the subject's ability to comply with the protocol.
* Active Hepatitis B virus infections
* Severe tremor/ataxia of the UE as defined by an EDSS with Cerebellar Functional System score of 3 or more due to upper extremity score (moderate tremor or clumsy movements interfere with function in all spheres)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in a clinical setting for the treatment of Multiple Sclerosis who are interested in starting Ocrevus but who are currently not on Ocrevus
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Y Maldonado, MD, Principal Investigator — University of South Florida
Locations (1):
- Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamers I, Feys P. Assessing upper limb function in multiple sclerosis. Mult Scler. 2014 Jun;20(7):775-84. doi: 10.1177/1352458514525677. Epub 2014 Mar 24. PMID 24664300
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Ontaneda D, Fox RJ, Chataway J. Clinical trials in progressive multiple sclerosis: lessons learned and future perspectives. Lancet Neurol. 2015 Feb;14(2):208-23. doi: 10.1016/S1474-4422(14)70264-9. PMID 25772899
- [Background] Schwid SR, Goodman AD, McDermott MP, Bever CF, Cook SD. Quantitative functional measures in MS: what is a reliable change? Neurology. 2002 Apr 23;58(8):1294-6. doi: 10.1212/wnl.58.8.1294. PMID 11971105
- [Background] Hamilton GF, McDonald C, Chenier TC. Measurement of grip strength: validity and reliability of the sphygmomanometer and jamar grip dynamometer. J Orthop Sports Phys Ther. 1992;16(5):215-9. doi: 10.2519/jospt.1992.16.5.215. PMID 18796752
- [Background] Benedict RH, Holtzer R, Motl RW, Foley FW, Kaur S, Hojnacki D, Weinstock-Guttman B. Upper and lower extremity motor function and cognitive impairment in multiple sclerosis. J Int Neuropsychol Soc. 2011 Jul;17(4):643-53. doi: 10.1017/S1355617711000403. PMID 21486517
- [Background] Stratford P, Binkley J, Stratford D. Development and initial validation of the upper extremity functional index. Physiotherapy Canada 2001;53(4):259-67.
- [Background] Ropper AH, Samuels M.A. Principals of Neurology. 9th edition. New York: McGraw-Hill, 2009.
- [Background] Genentech. Ocrevus™: Highlights of prescribing information. 2017.
- [Background] Goodin DS. Multiple Sclerosis and Related Disorders. Amsterdam, The Netherlands: Elsevier, 2014.
- [Background] Fox, EJ, Markowitz, C, Montalban, X, et al. Effect of Ocrelizumab on Upper Extremity Function in Patients With Primary Progressive Multiple Sclerosis in the ORATORIO Study. Presented at the 7th Joint European Committee for Treatment and Research in Multiple Sclerosis (ECTRIMS) and Americas Committee for Treatment and Research in Multiple Sclerosis (ACTRIMS) Meeting; 25-28 October 2017; Paris, France.
- [Result] Montalban X, Hauser SL, Kappos L, Arnold DL, Bar-Or A, Comi G, de Seze J, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Rammohan KW, Selmaj K, Traboulsee A, Sauter A, Masterman D, Fontoura P, Belachew S, Garren H, Mairon N, Chin P, Wolinsky JS; ORATORIO Clinical Investigators. Ocrelizumab versus Placebo in Primary Progressive Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):209-220. doi: 10.1056/NEJMoa1606468. Epub 2016 Dec 21. PMID 28002688
- [Result] Hauser SL, Bar-Or A, Comi G, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Montalban X, Rammohan KW, Selmaj K, Traboulsee A, Wolinsky JS, Arnold DL, Klingelschmitt G, Masterman D, Fontoura P, Belachew S, Chin P, Mairon N, Garren H, Kappos L; OPERA I and OPERA II Clinical Investigators. Ocrelizumab versus Interferon Beta-1a in Relapsing Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):221-234. doi: 10.1056/NEJMoa1601277. Epub 2016 Dec 21. PMID 28002679
- [Result] Cohen JA, Cutter GR, Fischer JS, Goodman AD, Heidenreich FR, Jak AJ, Kniker JE, Kooijmans MF, Lull JM, Sandrock AW, Simon JH, Simonian NA, Whitaker JN. Use of the multiple sclerosis functional composite as an outcome measure in a phase 3 clinical trial. Arch Neurol. 2001 Jun;58(6):961-7. doi: 10.1001/archneur.58.6.961. PMID 11405811
- [Result] Lamers I, Kelchtermans S, Baert I, Feys P. Upper limb assessment in multiple sclerosis: a systematic review of outcome measures and their psychometric properties. Arch Phys Med Rehabil. 2014 Jun;95(6):1184-200. doi: 10.1016/j.apmr.2014.02.023. Epub 2014 Mar 13. PMID 24631802
- [Result] Feys P, Duportail M, Kos D, Van Asch P, Ketelaer P. Validity of the TEMPA for the measurement of upper limb function in multiple sclerosis. Clin Rehabil. 2002 Mar;16(2):166-73. doi: 10.1191/0269215502cr471oa. PMID 11911515
- [Result] Gijbels D, Lamers I, Kerkhofs L, Alders G, Knippenberg E, Feys P. The Armeo Spring as training tool to improve upper limb functionality in multiple sclerosis: a pilot study. J Neuroeng Rehabil. 2011 Jan 24;8:5. doi: 10.1186/1743-0003-8-5. PMID 21261965
- [Result] Chesworth BM, Hamilton CB, Walton DM, Benoit M, Blake TA, Bredy H, Burns C, Chan L, Frey E, Gillies G, Gravelle T, Ho R, Holmes R, Lavallee RL, MacKinnon M, Merchant AJ, Sherman T, Spears K, Yardley D. Reliability and validity of two versions of the upper extremity functional index. Physiother Can. 2014 Summer;66(3):243-53. doi: 10.3138/ptc.2013-45. PMID 25125777
- [Result] Yozbatiran N, Baskurt F, Baskurt Z, Ozakbas S, Idiman E. Motor assessment of upper extremity function and its relation with fatigue, cognitive function and quality of life in multiple sclerosis patients. J Neurol Sci. 2006 Jul 15;246(1-2):117-22. doi: 10.1016/j.jns.2006.02.018. Epub 2006 May 5. PMID 16678208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occured July 2018 through September 2020 at a university medical clinic.
Groups:
- <20% Change of Clinical Stabalization From Baseline: This arm included patients who experienced <20% change in upper extremity function from baseline to 24 months.
Period: Overall Study
Arm/Group | <20% Change of Clinical Stabalization From Baseline
Started | 18
Completed | 15
Not Completed | 3
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Clinical Stabilization (Defined as no Significant Change (≤20%) From Baseline: Measure of upper extremity function over 24 months after initiation of Ocrevus™
Arm/Group | Clinical Stabilization (Defined as no Significant Change (≤20%) From Baseline
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Stabilization of Scores Using the Test d'Evaluation de la Performance Des Membres Supérieurs Des Personnes Agées (TEMPA) -Translasted in English to Mean "Performance Evaluation Test for the Elderly"
Description: The TEMPA is designed to assess the capabilities and limitations of upper limb function and consists of 9 tasks that mimic tasks of daily living that include picking up a jar, taking a spoonful of coffee from a jar, pouring water from a pitcher, handling coins, writing on an envelope and opening a pill container, tying a scarf around one's neck, shuffle and deal playing cards, and picking up and moving small objects. Each task is assessed by a rater by measuring speed of execution (seconds) and by functional rating of the subject's independence in performing them using an ordinal scale of 0 (completed without difficulty) to -3 (could not complete the task).
Time Frame: 24 months
Population: cohort of patients with Multiple Sclerosis from University of South Florida Multiple Sclerosis Center.
  Individuals, ages 18-70, with relapsing or progressive forms of MS and UE impairment that satisfied the approved indication for ocrelizumab and received ocrelizumab treatment commercially were assessed quarterly and semi-annually over 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | <20% Change of Clinical Stabalization From Baseline
Number analyzed (Participants) | 15
Participants | 12

2. Secondary Outcome: Stabilization of the Upper Extremity Functional Index (UEFI)
Description: The Upper Extremity Functional Index (UEFI) is a self-administered questionnaire which measures disability in patients with upper extremity conditions on a 5-point Likert scale. Scores range from 0 to 60 with lower scores indicating more functional difficulty in performing activities of daily living using the upper extremities including household and work activities, hobbies, lifting a bag of groceries, washing their scalp, pushing up on their hands, driving etc.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Stabilization (Defined as no Significant Change (≤20%) From Baseline
Number analyzed (Participants) | 14
Participants | 9

3. Secondary Outcome: Stabilization of 9-Hole Peg Test Scores
Description: The 9HPT is an objective measure of finger dexterity and upper extremity function, which is a widely used measure across most clinical trials in multiple sclerosis populations. The test involves the participant picking up and placing pegs one at time in the 9 holes and removing the pegs from their respective holes as quickly as possible. The participant completes the tasks twice on using their dominant hand, then twice on their non-dominant hand. Higher scores indicate a worse outcome.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Stabilization (Defined as no Significant Change (≤20%) From Baseline
Number analyzed (Participants) | 15
Participants | 11

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- <20% Change of Clinical Stabalization From Baseline: This arm included patients who experienced <20% in upper extremity function from baseline to 24 months.
Arm/Group | <20% Change of Clinical Stabalization From Baseline
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | <20% Change of Clinical Stabalization From Baseline (N=18)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Sepsis (Gastrointestinal disorders) | 1 (1)
Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | <20% Change of Clinical Stabalization From Baseline (N=18)
Urinary Tract Infection (Infections and infestations) | 5 (5)
Gradual Worsening of Trunk Strength (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Weakness of Right Hand (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased spasticity (Musculoskeletal and connective tissue disorders) | 2 (2)
Benign Prostatic Hyperplasia (Renal and urinary disorders) | 1 (1)
Falls (Musculoskeletal and connective tissue disorders) | 7 (8)
Bilateral Leg Edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Severe Fatigue (Endocrine disorders) | 1 (1)
Fatigue (Endocrine disorders) | 1 (1)
Increased Fatigue (Endocrine disorders) | 3 (3)
Increased spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased anxiety (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
right leg spasticity (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Bilateral Spasticity (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent Spasticity Increased (Abdomen to Knees) (Musculoskeletal and connective tissue disorders) | 1 (1)
right foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
mild pain due to fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Side Mid Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Painful Urination (Renal and urinary disorders) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Increased Right Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Itchy and Painful Throat (General disorders) | 1 (1)
Left Forearm Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral Ankle Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent Bilateral Calf Pain (Metabolism and nutrition disorders) | 1 (1)
Intermittent Bilateral Arm Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Difficulty Moving Right Leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased weakness right side of body (Nervous system disorders) | 1 (1)
MS Exacerbation Flare (Nervous system disorders) | 1 (1)
Broken Rib (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg Swelling (L foot, ankle, leg from knee down) (Musculoskeletal and connective tissue disorders) | 1 (1)
Weakness (Nervous system disorders) | 1 (1)
Lymphedema (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Loose Cough (Infections and infestations) | 1 (1)
Night Sweats (Infections and infestations) | 1 (1)
Asthma Exacerbation (Infections and infestations) | 1 (1)
Acute Hypoxic Respiratory Failure (Infections and infestations) | 1 (1)
Face and Head Numbness (Nervous system disorders) | 1 (1)
Acute Bronchitis (Infections and infestations) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 2 (2)
Worsening Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 1 (1)
Increased Left Left Numbness (Nervous system disorders) | 1 (1)
Intermittent Headaches (General disorders) | 3 (3)
Dry Skin Bilateral Lower Legs (Skin and subcutaneous tissue disorders) | 1 (1)
Decreased Balance (Nervous system disorders) | 3 (3)
Intermittent Itchiness of the Face (Skin and subcutaneous tissue disorders) | 1 (1)
Left Leg Burning Sensation (Nervous system disorders) | 1 (1)
Left Leg Spasms (Nervous system disorders) | 1 (1)
Worsening Whole Body Spasms (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Increased Bilateral Hand Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Leg Weakness Bilateral (Musculoskeletal and connective tissue disorders) | 1 (1)
Hair loss (General disorders) | 1 (1)
Increased Hair Loss (General disorders) | 1 (1)
Increased Bilateral Foot Numbness (Nervous system disorders) | 2 (2)
Increased Bilateral Hand Numbness (Nervous system disorders) | 1 (1)
Bilateral Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Increased Foot Drop (Nervous system disorders) | 1 (1)
Increased Right Foot Drop (Nervous system disorders) | 1 (1)
Memory Decline (General disorders) | 2 (2)
High Blood sugar (Blood and lymphatic system disorders) | 2 (2)
Cellulitis Foot (Infections and infestations) | 1 (1)
Dry Skin Patches on Hands and Back (Skin and subcutaneous tissue disorders) | 1 (1)
Infusion Related Reaction Formication (Nervous system disorders) | 1 (1)
Bilateral Small Red Blotches on Skin of Arms (Skin and subcutaneous tissue disorders) | 1 (1)
viral Infection (Infections and infestations) | 1 (1)
Increased Leg Weakness (Nervous system disorders) | 1 (1)
Increased Generalized Weakness (Nervous system disorders) | 1 (1)
Intermittent Vomiting (Gastrointestinal disorders) | 1 (1)
Abnormal Kidney Function (Hepatobiliary disorders) | 1 (1)
Increased Bilateral Leg Heaviness (General disorders) | 1 (1)
Bilateral Leg Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Arm Numbness (Nervous system disorders) | 1 (1)
Tricuspid Regurgitation (Cardiac disorders) | 1 (1)
Compound Melanocytic Nevus with Features of a Dysplastic Nevus of the Left Abdomen (Skin and subcutaneous tissue disorders) | 1 (1)
Worsening Essential Tremor Bilateral Hands (Nervous system disorders) | 1 (1)
Floater Left Eye (Eye disorders) | 1 (1)
Partial Detached Retina Left Eye (Eye disorders) | 1 (1)
Chronic Low Blood Pressure (General disorders) | 1 (1)
Worsening Arthritis Bilateral Hands (Musculoskeletal and connective tissue disorders) | 2 (2)
Sciatica Left Side (Nervous system disorders) | 1 (1)
Infusion Related Reaction: Itchy Throat (General disorders) | 1 (1)
Covid-19 vaccine (Surgical and medical procedures) | 1 (1)
Worsening Bilateral Hand Cramping (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Right Foot Drop (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth pulled (General disorders) | 1 (1)
Chronic Bilateral Leg Weakness (Nervous system disorders) | 1 (1)
Left Knee Small Cyst Growth (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Low Iron (Blood and lymphatic system disorders) | 1 (1)
High Cholesterol (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Drainage (Skin and subcutaneous tissue disorders) | 1 (1)
Intermittent Weakness (Nervous system disorders) | 1 (1)
Chronic Deep Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Infusion Related Reaction: Chronic Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tingling of Interglutal Cleft (Nervous system disorders) | 1 (1)
Numbness of Interglutal Cleft (Nervous system disorders) | 1 (1)
Right Knee Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Eye Cataract Surgery (Surgical and medical procedures) | 1 (1)
Mucosal Thickening Removal From Sinus Cavity (Surgical and medical procedures) | 1 (1)
Right Shoulder Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Covid-19 infection (Infections and infestations) | 1 (1)
Intermittent Migraines (General disorders) | 1 (1)
Increased Right Arm Tremors (Nervous system disorders) | 1 (1)
Increased Bilateral Hand Tremors (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03562975/Prot_SAP_000.pdf